CLINICAL TRIAL: NCT00182988
Title: Alzheimer's Caregiver Ratings of Communication & Coping Behavior
Brief Title: Alzheimer's Caregiver Communication Study
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Pamela A. Saunders, Ph.D., Georgetown University
Other Study IDs: IA0082; 1R03AG022627 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Alzheimer's Disease
Keywords: communication behavior; coping; functional ability; quality of life; caregiving
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The point of this research is to improve the communicative relationship between the caregiver and care receiver. It is input from the caregiver on these communicative behaviors that will inform the process of understanding how to reduce the caregiver burden that comes from this communicative relationship.

DETAILED DESCRIPTION:
This research study is developing a new checklist to measure communicative coping behaviors of persons with Alzheimer's Disease in the home environment. The Communicative Coping Behavior Checklist (CCBC) is an observation checklist to be completed by the caregiver or knowledgeable informant. The current version includes 23 behaviors to be rated for frequency and effectiveness. The behaviors that will be observed cover management of memory loss within three broad categories: humor, explanations, and general coping behaviors.

Two kinds of couples will participate in this study. One includes a person with Alzheimer's Disease and their caregiver. The second includes a cognitively intact participant and study partner, both over the age of 60, to serve as controls.

Study Visit 1 (3 hours long) During the first visit, the person with Alzheimer's Disease/control participant can expect to be asked questions about their memory, thinking and concentration, demographics, quality of life, and mood. The caregiver/study partner will be asked about their quality of life, mood, and daily activities.

At the end of the visit the caregiver/study partner will be given a copy of the CCBC and asked to take it home. S/he will be instructed to rate the person with Alzheimer's Disease/ control participant's communicative coping behavior over the course of the next two weeks. At the end of that time, a research assistant will call the caregiver/study partner and administer the CCBC over the telephone.

Study Visit 2 (3 hours long) The second visit will occur in the clinic approximately 12 months from the date of the first visit. As with the first study visit, again both the person with Alzheimer's Disease/control participant and the caregiver/study partner will answer questions about their memory, quality of life, mood, and daily activities. Once again, the caregiver/study partner will be given a copy of the CCBC and asked to take it home and complete.

Both visits will take about three hours for the caregiver/study partner and about two hours for the person with dementia or control subject.

ELIGIBILITY:
*Note* Currently enrolling participants for control group only

Inclusion Criteria:

* Couples including spouse or family member who spend at least 2-3 hours per day together
* Both must be cognitively intact

Exclusion Criteria:

* Cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2004-10; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Saunders, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States